CLINICAL TRIAL: NCT01989988
Title: A Randomized Trial Study of Different Laparoscopic Gastric Bypass Surgery in Patients With Obesity-related T2DM
Brief Title: DMBSS-A Randomized Trial of Different Laparoscopic Gastric Bypass Surgery in Patients With Obesity-related T2DM
Acronym: DMBSS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Min-Sheng General Hospital (Other)
Responsible Party: Principal Investigator, WEI-CHENG YAO, Department of Surgery, Min-Sheng General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MSIRB2013003; MSIRB2013003 (Other: MSIRB)
Record Dates: First submitted 2013-01-22; First posted 2013-11-21 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Diabetes Mellitus Type 2 in Obese
Keywords: Type 2 Diabetes Mellitus (T2DM); Obesity; Laparoscopic gastric bypass; Duodenum exclusion
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- LRYGB (Active Comparator): 20 subjects Randomized will undergo LRYGB surgery
  Interventions: Procedure: LRYGB
- SADJB (Active Comparator): 20 subjects will undergo SADJB surgery
  Interventions: Procedure: SADJB
- LMGB (Active Comparator): 20 subjects will undergo LMGB surgery
  Interventions: Procedure: LMGB

INTERVENTIONS:
Procedure: LMGB
  Arms: LMGB
Procedure: LRYGB
  Arms: LRYGB
Procedure: SADJB
  Arms: SADJB

SUMMARY:
The investigators would like to conduct a randomized clinical trial to compare the efficacy of diabetes treatment between different gastric bypass procedures involving type 2 diabetics patients with BMI from 27.5 to 35 kg/m2

DETAILED DESCRIPTION:
The investigators would like to conduct a randomized clinical trial to compare the efficacy of diabetes treatment between different gastric bypass procedures involving type 2 diabetics patients with BMI from 27.5 to 35 kg/m2. This program will determine the relative effectiveness among LMGB 、RYGB and SADJB .The primary end point including HbA1C<6.0%, LDL-C<100mg/dl and SBP<130mmHg at one year after surgery. Through this study, the investigators may understand which gastric bypass is the best for type 2 diabetic's treatment. The investigators also hope some new treatment modulation may be developed.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 to 67 years
* Diagnosed with T2DM at least 6 months prior to enrollment, under the active care of a doctor for at least the six months prior to enrollment, HbA1c ≥ 7.5 %
* Body Mass Index (BMI) ≥ 27.5 kg/m 2 and ≤ 34.9 kg/m 2
* Willingness to accept random assignment to either treatment group.
* Willingness to comply with the follow-up protocol
* Written informed consent.

Exclusion Criteria:

* Cardiovascular event (myocardial infarction, acute coronary syndrome, coronary artery angioplasty or bypass, stroke) in the past six months.
* Current evidence of congestive heart failure, angina pectoris, or symptomatic peripheral vascular disease.
* Cardiac stress test indicating that surgery would not be safe.
* Pulmonary embolus or thrombophlebitis in the past six months
* Cancer of any kind (except basal cell skin cancer or cancer in situ) unless documented to be disease-free for five years
* Serum creatinine ≥ 1.5 mg/dl
* History of stomach surgery, bile duct surgery, pancreatic surgery, splenectomy, or colon resection
* Previous organ transplantation.
* History of alcohol or drug dependency
* Current participation in a conflicting research protocol.

Ages: 20 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-07 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Remission of diabetes | two years
  remission of Diabetes Mellitus Type 2 after different types of Gastric bypass surgery

SECONDARY OUTCOMES:
weight loss and improvement in quality of life | 2 years
  weight loss and improvements in quality of life after different types of gastric bypass surgery

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Jei Lee, M.D., PH.D, Study Chair — Min-Sheng General Hospital
Locations (1):
- Min-Sheng General Hospital, Taoyuan, Taiwan